CLINICAL TRIAL: NCT02539927
Title: International Multicentre Validation Study of SAGIT® Instrument in Acromegaly
Brief Title: Validation Study of the SAGIT® Instrument in Acromegaly
Acronym: SAGIT
Status: Completed | Type: Observational
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Other Study IDs: 8-79-52030-295
Record Dates: First submitted 2015-07-07; First posted 2015-09-03 (Estimated); Last update posted 2018-11-01 (Actual); Status verified 2018-10

CONDITIONS: Acromegaly
MeSH Terms: conditions — Acromegaly

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Controlled
- Not controlled
- Control status yet to be clarified

SUMMARY:
Patients will be treated in accordance with the standard medical practice of the hospital where they have been recruited during their participation in this study. No additional assessments or tests will be required.

SAGIT® is a new instrument developed by a group of acromegaly experts to help practicing endocrinologists to manage acromegalic patients and disease activity in their clinical practice and define acromegaly staging. It reports 5 elements: Signs and symptoms - S; Associated comorbidities - A; Growth hormone (GH) concentration - G; Insulin-like growth factor 1(IGF-1) concentration -I; Tumour size- T.

The instrument has been pre evaluated during a qualitative pilot study. The purpose of the validation study is to define and validate the scoring of the SAGIT® instrument.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18 years-old or above at study inclusion
* Treatment-naïve and non treatment-naïve patients with a diagnosis of acromegaly
* Data required to complete the SAGIT® tool are available in the patient medical records and do not require additional assessments or tests
* Data required to complete the SAGIT® tool are recorded within the 3 months preceding the inclusion visit (6 months for MRI)

Exclusion Criteria:

* Acute uncontrolled disease requiring intensive care

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients suffering from Acromegaly in specialist care clinics and hospital clinics.
Sampling Method: Non-Probability Sample
Enrollment: 227 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2018-09-03 (Actual); Study Completion 2018-09-03 (Actual)

PRIMARY OUTCOMES:
Define and validate the scoring of the SAGIT® instrument | baseline
  Evaluating the ability of the instrument to discriminate subgroups of subjects with acromegaly (controlled vs not controlled).

SECONDARY OUTCOMES:
The ability of the SAGIT® instrument to predict the occurrence of significant clinical event(s) and/or treatment change(s) over time. | 2 years
  Significant clinical event is defined as death, stroke, onset of diabetes, onset of arthritis/onset of arthritis disability, myocardial infarction and/or diagnosis of other tumor; treatment change is defined as change in therapeutic doses, in therapeutic drug class, surgery or radiotherapy.
Define SAGIT® characteristics for different groups | 2 years
  Controlled vs. non controlled. Treatment-naïve, patients vs. currently treated vs. previously treated patients
The association between the SAGIT® tool and patients' quality of life measured using Acromegaly Quality of Life (AcroQoL) scores. | 2 years
  Acromegaly Quality of Life (AcroQoL) scores will be compared between patient groups defined according to SAGIT scoring algorithm (controlled vs. not controlled). This comparison will be performed using t-tests for each available visit of the prospective population.

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (32):
- United States (4):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - The Emory Pituitary Center, Atlanta, Georgia
  - Cleveland Clinic, Cleveland, Ohio
  - Endocrinology and Metabolism, Pittsburgh, Pennsylvania
- CHU de Liège, Liège, Belgium
- Brazil (2):
  - Federal University of Rio de Janeiro, Rio de Janeiro
  - University Hospital, São Paulo
- Denmark (2):
  - Department of Clinical Medicine - The Department of Endocrinology and Diabetes, Aarhus C
  - University Hospital, Dept of Endocrinology, Copenhagen
- France (4):
  - Hopital Neuro-Cardiologique, Bron
  - Hopital de Bicêtre, Le Kremlin-Bicêtre
  - CHU de Marseille - Hôpital de la Timone, Marseille
  - CHU Larrey, Toulouse
- Germany (3):
  - University Hospital, Essen
  - Endoc Zentrum Fûr Endokrine Tumoren, Hamburg
  - Private Clinique, Oldenburg
- Italy (5):
  - Ospedaliera Spedali Civili di Brescia, Montichiari
  - Azienda Ospedaliero Universitar a Fedderico II, Naples
  - Azienda Ospedaliera di Padova, Padua
  - Azienda Ospedaliero Universitaria Pisana-Endcrinologia 2, Pisa
  - Endocrinology, University Hospital, Policlinica Gemelu, Rome
- Netherlands (3):
  - LUMC Leiden,, Leiden
  - Radbound UMC, Nijmegen
  - Erasmus MC, Rotterdam
- Spain (4):
  - University Hospital, Barcelona
  - University Hospital, Madrid
  - Hospital de Condia(CHUS) RVA Ramon Baltar S/N, Santiago de Compostela
  - University Hospital Virgen del Rocio, Seville
- United Kingdom (4):
  - Aberdeen Royal Infirmary, Aberdeen
  - University Hospital, Cambridge
  - Université Hospital, Cardiff
  - Endocrinology and Metabolism Churchill Hospital, Oxford

REFERENCES:
- [Derived] Giustina A, Bronstein MD, Chanson P, Petersenn S, Casanueva FF, Sert C, Houchard A, Melmed S. International Multicenter Validation Study of the SAGIT(R) Instrument in Acromegaly. J Clin Endocrinol Metab. 2021 Nov 19;106(12):3555-3568. doi: 10.1210/clinem/dgab536. PMID 34313752
- [Derived] Giustina A, Bronstein MD, Chanson P, Petersenn S, Casanueva FF, Sert C, Houchard A, Melmed S. Staging and managing patients with acromegaly in clinical practice: baseline data from the SAGIT(R) validation study. Pituitary. 2019 Oct;22(5):476-487. doi: 10.1007/s11102-019-00977-5. PMID 31338660